CLINICAL TRIAL: NCT01705236
Title: A 3-year Multi-center Study to Describe the Long Term Changes of Optical Coherence Tomography (OCT) Parameters in Patients Under Treatment With Gilenya®
Brief Title: A 3-year Multi-center Study to Describe Changes of OCT Parameters Under Treatment With Gilenya®
Acronym: PASSOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CFTY720DDE15TS
Record Dates: First submitted 2012-08-13; First posted 2012-10-12 (Estimated); Results first posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis RRMS
Keywords: Multiple sclerosis (MS); MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fingolimod - Longitudinal Assessment (Experimental): No study drug was provided. Fingolimod was to be prescribed according to local label. The decision to prescribe fingolimod had to be made independent of this study.
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod — All subjects received an oral dose of 0.5 mg fingolimod (FTY720) per capsule (hard gelatin capsules) once daily according to local label for the treatment of their MS.
  Other Names: FTY720

SUMMARY:
This was a 3-year, prospective, multi-center, open-label study to describe the long term changes of optical coherence tomography (OCT) parameters in RRMS patients under treatment with Fingolimod. It was designed to longitudinally study the degeneration of retinal axons by measuring change in RNFL thickness by latest OCT-technology.

ELIGIBILITY:
Inclusion Criteria

Patients eligible for inclusion in this study have to fulfill all of the following criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Male or female subjects aged 18-65 years.
3. Subjects with relapsing remitting MS defined by 2010 revised McDonald criteria (see Appendix 4).
4. Patients with Expanded Disability Status Scale (EDSS) score of 0-6.0 inclusive (see Appendix 6).
5. Patients stable on immunomodulatory treatment with fingolimod for at least 1 month and at most 4 months prior to screening according to local label
6. Neurologically stable with no evidence of relapse within 30 days prior to inclusion date
7. Sufficient ability to read, write, communicate and understand

Exclusion Criteria

Patients fulfilling any of the following criteria are not eligible for inclusion in this study:

1. Patients who have been treated with:

   * systemic corticosteroids or immunoglobulins within 1 month prior to screening;
   * immunosuppressive medications such as azathioprine, cyclophosphamide, or methotrexate within 3 months prior to screening;
   * monoclonal antibodies (including natalizumab) within 3 months prior to screening;
   * mitoxantrone within 6 months prior to screening
   * cladribine at any time.
2. Patients with any medically unstable condition, as assessed by the primary treating physician at each site.
3. Patients with any of the following cardiovascular conditions :

   * history of myocardial infarction or with current unstable ischemic heart disease;
   * Heart failure (NYHA III-IV) or any severe cardiac disease as determined by the Investigator (see Appendix 5);
   * history or presence of a second-degree AV block, Type II or a third-degree AV block
   * patients receiving Class Ia (ajmaline, disopyramide, procainamide, quinidine) or III antiarrhythmic drugs (e.g., amiodarone, bretylium, sotalol, ibulitide, azimilide, dofelitide);
   * proven history of sick sinus syndrome;
   * uncontrolled hypertension
4. Patients with severe respiratory disease, pulmonary fibrosis, or chronic obstructive pulmonary disease (Class III-IV).
5. Patients with history of specific MRI findings (tumor, subdural haematoma, post-contusional changes, territorial stroke, neurodegenerative disorders, aneurysm/arteriovenous malformation, evidence of past macroscopic haemorrhage, or other relevant MRI findings that would interfere with evaluation)
6. Any severe disability or clinical impairment that can prevent the patient to meet all study requirements at the investigator's discretion
7. History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin
8. Patients who have received an investigational drug (excluding fingolimod) or therapy within 90 days or 5 half-lives of screening, whichever is longer.
9. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG test (serum)
10. Patients with any ophthalmologic reason for RNFL pathology other than MS, such as: optic neuropathy, active advanced glaucoma, injury of the optic nerve based on the ophthalmologist's clinical judgment
11. history or presence of severe myopia

    1. in patients who have not had refractive surgery, a refractive error of greater than 6.00 diopters
    2. pathologic fundus changes of high myopia, such as retinal pigmentary atrophy, besides peripapillary atrophy (atrophy involving the macula) or a staphyloma
    3. in patients that have had previous refractive surgery, an axial eye length of greater than 26 mm
12. Acute optic neuritis within the past 6 months before screening
13. Evidence of advanced, non-proliferative or proliferative diabetic retinopathy
14. Presence of retinal conditions associated with edema, subretinal fluid, cysts, etc.
15. Concomitant use of drugs that may directly affect retinal structure and function (e.g.

chronic systemic corticosteroids [>30 consecutive days; doses higher than Cushing threshold e.g. prednisone 7.5mg/d], intraocular anti-angiogenic drugs [ranibizumab, bevacizumab], intraocular steroids etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-08-20 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- Germany (9):
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened at 10 study centers in Germany (9 centers) and Switzerland (1 center).
Pre-assignment Details: Subjects who passed the screening were enrolled in the trial.
Groups:
- Fingolimod - Longitudinal Assessment: No study drug was provided. Fingolimod was to be prescribed according to local label. The decision to prescribe fingolimod was to be made independent of this study.
Period: Overall Study
Arm/Group | Fingolimod - Longitudinal Assessment
Started | 87
Completed | 60
Not Completed | 27
Not completed — Lost to Follow-up | 1
Not completed — Administrative problems | 2
Not completed — Unsatisfactory therapeutic effect | 3
Not completed — Protocol Violation | 3
Not completed — Abnormal test procedure result(s) | 4
Not completed — Abnormal laboratory value(s) | 4
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Arm/Group | Fingolimod - Longitudinal Assessment
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 84
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 36 in Average Retinal Nerve Fiber Layer Thickness (RNFLT)
Description: The primary endpoint was the change, i.e. the absolute difference, in average RNFL thickness from baseline to month 36 (or last values in case of missing data) in the Full Analysis Set (FAS). Average RNFL thickness was the average of valid measurements of the right and left eye and assessed by optical coherence tomography (OCT).
Time Frame: Baseline, month 36
Population: Full Analysis Set (FAS). The FAS consisted of all subjects treated with fingolimod who had at least one post-baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Fingolimod - Longitudinal Assessment
Number analyzed (Participants) | 72
micrometer | -1.5 (2.7)

2. Secondary Outcome: Change From Baseline to Month 12 and 24 in Average Retinal Nerve Fiber Layer Thickness (RNFLT)
Description: Change from baseline in average RNFL thickness to months 12 and 24 (or last values in case of missing data) in the Full Analysis Set (FAS). Average RNFL thickness was the average of valid measurements of the right and left eye and assessed by optical coherence tomography (OCT).
Time Frame: Baseline, month 12, month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Fingolimod - Longitudinal Assessment
Number analyzed (Participants) | 72
micrometer
  Change from baseline to month 12 | -0.8 (2.4)
  Change from baseline to month 24 | -1.1 (2.4)

3. Secondary Outcome: Change From Baseline to Month 12, 24 and 36 in Average Quadrant Retinal Nerve Fiber Layer Thickness (RNFLT)
Description: Change from baseline in average quadrant RNFL thickness to months 12, 24 and 36 (or last values in case of missing data) in the Full Analysis Set (FAS). Average quadrant RNFL thickness was the average of valid measurements of the right and left eye and assessed by optical coherence tomography (OCT). Quadrant RNFL thickness were: Nasal-inferior; nasal-superior; temporal-inferior; temporal-superior.
Time Frame: Baseline, month 12, month 24, month 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Fingolimod - Longitudinal Assessment
Number analyzed (Participants) | 72
micrometer
  Nasal-superior RNFL thickness: month 12 | 0.5 (4.0)
  Nasal-superior RNFL thickness: month 24 | -0.4 (3.4)
  Nasal-superior RNFL thickness: month 36 | -0.7 (3.9)
  Nasal-inferior RNFL thickness: month 12 | -1.2 (4.9)
  Nasal-inferior RNFL thickness: month 24 | -1.6 (5.1)
  Nasal-inferior RNFL thickness: month 36 | -2.1 (5.2)
  Temporal-inferior RNFL thickness: month 12 | -1.2 (2.5)
  Temporal-inferior RNFL thickness: month 24 | -1.6 (3.1)
  Temporal-inferior RNFL thickness: month 36 | -2.3 (4.1)
  Temporal-superior RNFL thickness: month 12 | -0.5 (3.9)
  Temporal-superior RNFL thickness: month 24 | -0.4 (3.4)
  Temporal-superior RNFL thickness: month 36 | -1.1 (4.1)

4. Secondary Outcome: Change From Baseline to Month 12, 24 and 36 in Total Macular Volume (TMV)
Description: Change from baseline in TMV to months 12, 24 and 36 (or last values in case of missing data) in the Full Analysis Set (FAS).
Time Frame: 12, 24 and 36 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cubic millimeter
Arm/Group | Fingolimod - Longitudinal Assessment
Number analyzed (Participants) | 72
Cubic millimeter
  Change from baseline to month 12: number analyzed (Participants) | 71
  Change from baseline to month 12 | -0.03 (0.08)
  Change from baseline to month 24: number analyzed (Participants) | 71
  Change from baseline to month 24 | -0.04 (0.08)
  Change from baseline to month 36: number analyzed (Participants) | 71
  Change from baseline to month 36 | -0.06 (0.10)

5. Secondary Outcome: Change From Baseline to Month 12, 24 and 36 in Ganglion Cell Inner Plexiform (GCIP)
Description: Change from baseline in GCIP to months 12, 24 and 36 (or last values in case of missing data) in the Full Analysis Set (FAS).
  The change in Ganglion cell layer thickness (GCLT) had been defined as secondary endpoint in the protocol, but OCT measured the GCIP instead. This was done because both layers were not clearly separable by OCT. GCIP was calculated as mean of the inner sectors (nasal, superior, temporal, and inferior) and declared as usual parameter instead. This change was introduced prior to data base lock, but the derivation of GCIP was corrected after data base lock.
Time Frame: Baseline, month 12, month 24, month 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Fingolimod - Longitudinal Assessment
Number analyzed (Participants) | 72
micrometer
  Change from baseline to month 12: number analyzed (Participants) | 71
  Change from baseline to month 12 | -0.49 (2.39)
  Change from baseline to month 24: number analyzed (Participants) | 71
  Change from baseline to month 24 | -0.42 (2.74)
  Change from baseline to month 36: number analyzed (Participants) | 71
  Change from baseline to month 36 | -0.46 (3.01)

6. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with adverse events and specifically macular edema.
Time Frame: 36 months
Population: Safety Population (SAF). The SAF consisted of all subjects treated with fingolimod for whom safety information had been collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Fingolimod - Longitudinal Assessment
Number analyzed (Participants) | 87
Participants
  No. of subjects with any AE | 80
  No. of subjects with macular edema | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment up to maximum duration of 36 months
Arm/Group | Fingolimod - Longitudinal Assessment
All-Cause Mortality (participants affected / at risk) | 0/87
Serious Adverse Events (participants affected / at risk) | 11/87
Other Adverse Events (participants affected / at risk) | 68/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod - Longitudinal Assessment (N=87)
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 1
ERYSIPELAS (Infections and infestations) | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 1
OPHTHALMIC HERPES ZOSTER (Infections and infestations) | 1
WOUND INFECTION (Infections and infestations) | 1
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1
SUTURE RELATED COMPLICATION (Injury, poisoning and procedural complications) | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1
CERVIX CARCINOMA STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
NASAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 2
NEURALGIC AMYOTROPHY (Nervous system disorders) | 1
UHTHOFF'S PHENOMENON (Nervous system disorders) | 1
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod - Longitudinal Assessment (N=87)
LYMPHOPENIA (Blood and lymphatic system disorders) | 9
DIARRHOEA (Gastrointestinal disorders) | 6
BRONCHITIS (Infections and infestations) | 6
CONJUNCTIVITIS (Infections and infestations) | 5
NASOPHARYNGITIS (Infections and infestations) | 41
SINUSITIS (Infections and infestations) | 6
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7
URINARY TRACT INFECTION (Infections and infestations) | 7
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 8
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7
DIZZINESS (Nervous system disorders) | 5
HEADACHE (Nervous system disorders) | 10
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 21
PARAESTHESIA (Nervous system disorders) | 5
DEPRESSION (Psychiatric disorders) | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 6
ALOPECIA (Skin and subcutaneous tissue disorders) | 5
HYPERTENSION (Vascular disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-03-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT01705236/SAP_000.pdf
  • Study Protocol (2016-07-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT01705236/Prot_001.pdf